CLINICAL TRIAL: NCT01106729
Title: Tracing the Path of the Plant Pigment Cyanidin-3-glucoside, Through the Human Body After Consumption
Brief Title: Tracing the Path of an Ingested Plant Pigment Through the Human Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Quadram Institute Bioscience (Other)
Responsible Party: Colin Kay, Chief Investigator, University of East Anglia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BB/H004963/1; R17228 (Other: University of East Anglia)
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Metabolism and Clearance of Cyanidin 3 Glucoside
Keywords: Flavonoids; Anthocyanin; Cyanidin 3 glucoside; Acute feeding trial; Stable isotope; Metabolism; Clearance; Bioavailability; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyanidin 3 glucoside (Other)
  Interventions: Dietary Supplement: Cyanidin 3 glucoside

INTERVENTIONS:
Dietary Supplement: Cyanidin 3 glucoside — Ingestion of 500mg of Cyanidin 3 glucoside (a naturally occurring plant pigment)

SUMMARY:
This study will trace the path of a natural plant pigment, (cyanidin-3-glucoside; C3G), through the human body after consumption. C3G is the most abundant of the naturally occurring anthocyanin family of plant pigments and is responsible for the red to purple colour of many fruits and vegetables. Anthocyanins are promoted as being potentially beneficial to heart-health and also have anti-cancer properties, however little is known about how the body processes these compounds after they are eaten or how they are cleared from the digestive system. The investigators study aims to answer these questions and, in doing so, unravel how they may benefit everyone's health.

In this BBSRC funded study, 8 healthy (18-45y) male participants will be recruited to a one day feeding study (lasting 8 hours) to establish the routes of clearance of anthocyanins from the body. After consent has been obtained, participants will be screened to establish their health (by NHS clinical staff). Eligible participants will be asked to consume a low anthocyanin diet for 7 days and to attend a study day at the Clinical Research & Trials Unit (CRTU, University of East Anglia). Participants will attend in a fasted state (at least 8h of water only) and will be asked to provide a urine (total morning void) and faecal (within the previous 72h) sample. Participants will then consume a C3G capsule and blood and breath samples will be collected at regular intervals after consumption (0.5, 1, 2, 4 and 6 hours). The capsule is roughly the size of a commercial vitamin-C tablet (500mg). Participants will then return in a fasted state on the following 2 mornings to provide further urine, faeces, breath and blood samples. Low anthocyanin meals will be provided throughout the study day and on the following 2 mornings. Participants will be reimbursed for their inconvenience

ELIGIBILITY:
Inclusion Criteria:

* Males
* 18-45 years old
* No allergies to fruits or vegetables containing anthocyanins or foods to be provided on the study day
* Those agreeing to restrict dietary intake of rich sources of anthocyanins
* Those agreeing to comply with a biological sampling protocol and have cannula inserted for the collection of blood samples on the study day
* Those agreeing to record their dietary intake over 3 days (1 weekend day and 2 week days)

Exclusion Criteria:

* Those judged by the study clinical staff (to be appointed) to have biochemical and / or haematological screening results which reflect compromised health or that may affect the study analysis
* Participants with a body mass index of less than 18.5 or greater than 30
* Taking food / dietary supplements containing anthocyanins e.g. grape seed extract, acai berry (unless prepared to cease intake during, and 7 days preceding the study)
* Parallel participation in another research project which involves dietary intervention and/or sampling of biological fluids/material
* Smokers or those who have ceased smoking within 12 months.
* Habitual drinkers of more than 4 units* of alcohol per day or more than 21 units per week (NHS guidelines). *A unit of alcohol is approximately equivalent to a half pint of full strength beer or cider or a small glass of wine (100ml) or a single measure (25ml) of spirits
* Having donated blood in the last month

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The outcome measure for this study is the measure of the total amount of the 'heavy' label (which was incorporated into the C3G) in the blood, urine, faeces and breath samples in the 48 hours following consumption. | 72 hours

SECONDARY OUTCOMES:
The secondary outcome measures is to identify the metabolites of C3G and the tertiary outcome measure is to establish the rates of clearance of both the heavy label and the identified metabolites. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Colin Kay, PhD, Principal Investigator — University of East Anglia; Charles Czank, PhD, Study Director — University of East Anglia; Aedin Cassidy, PhD, Study Director — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Czank C, Cassidy A, Zhang Q, Morrison DJ, Preston T, Kroon PA, Botting NP, Kay CD. Human metabolism and elimination of the anthocyanin, cyanidin-3-glucoside: a (13)C-tracer study. Am J Clin Nutr. 2013 May;97(5):995-1003. doi: 10.3945/ajcn.112.049247. PMID 23604435